CLINICAL TRIAL: NCT04056663
Title: Health-circuit Evaluation as a Digital Support for the Management of Patients at Risk of Hospitalization
Acronym: Health_Circuit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Carmen Herranz, Nurse, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Health-Circuit Clinic
Record Dates: First submitted 2019-07-22; First posted 2019-08-14 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Multiple Chronic Conditions; Chronic Disease
Keywords: Artificial Intelligence; Continuity of Patient Care
MeSH Terms: conditions — Multiple Chronic Conditions; Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health-Circuit mobile application (Experimental): The intervention contemplates. (i) management of unexpected events; and, (ii) empowering the patient to improve self-efficacy.
  Users of the intervention arm will have the Health-Circuit mobile application, which will offer them the possibility of contacting the case managers to notify a health event at any time and that this can be resolved by their health professionals through Health -Circuit. The improvement of the patient's self-efficacy for the management of their health problems through the use of Health-Circuit is considered through the virtual visits of follow-up with the manager, the possibility of interacting with the manager and the consultation of the shared documents reminders of the action plan agreed with the patient.
  Interventions: Behavioral: Health-Circuit mobile application
- Conventional treatment (No Intervention): Patients assigned to this group will follow conventional treatment. Once the three months have passed, we will contact you again to ask the pertinent questions.

INTERVENTIONS:
Behavioral: Health-Circuit mobile application — Health-Circuit as a collaborative tool between professionals and patient and professionals
  Arms: Health-Circuit mobile application

SUMMARY:
Background - There is a high potential for hospitalization prevention through: (i) a greater continuity of care, achieved by facilitating collaborative work among professionals at different levels of care, and (ii) improving the self-efficacy of patients. For both objectives, the support of appropriate information and communication technologies is essential. The study raises the hypothesis that an industry 4.0 system, Health-Circuit, based on communication technologies and intelligent collaboration, will facilitate a greater continuity of care and an improvement in patients' self-efficacy.

Objective - Analysis of Health-Circuit's potential for improving the continuity of care and self-efficacy of chronic patients at risk of hospitalization.

Material and methods - Controlled, single-blinded, randomized trial by primary care teams, with a 2:1 intervention-control ratio. The first phase of the study (September-November 2019) will be carried out in 75 patients from the primary care area of Barcelona Esquerra under the influence of Hospital Clínic of Barcelona (CAPSBE, 110k inhabitants). In the intervention group, the patients, and the corresponding healthcare professionals, will communicate and collaborate though Health-Circuit, while the control group will receive conventional treatment. In a second phase (beginning December 2019), the study will be extended to the entire healthcare area of Barcelona Esquerra (AISBE, 520k inhabitants).

Expected results - From a clinical perspective, a reduction in the number of urgent face-to-face visits is expected at: (i) Hospital; (ii) Primary Care, or, (iii) Primary Care Emergency Centers, due to better continuity of care and greater self-efficacy of patients. However, the results sought in Phase I of the study will be, fundamentally: (i) the evaluation of the usability and acceptability of Health-Circuit for patients and professionals, and (ii) the analysis of the potential of the digital tool for the management of complex clinical processes with the help of intelligent bots. In phase II of the study, the central objectives will be (i) increase in the capacity to resolve events, and (ii) improvement of patients' self-efficacy.

DETAILED DESCRIPTION:
The present investigation develops in the framework of the EU project CONNECARE "Personalized Connected Care for Complex Chronic Patients (H2020 - BHC25 - 689802), whose registration number in the medical research ethics committee of Hospital Clínic of Barcelona is HCB / 2018/0803. CONNECARE assumes that (i) the improvement of the continuity of care, associated with facilitating collaborative work among professionals of different levels of care, and, (ii) the increase in patients' self-efficacy, results in an optimization of the management of chronic patients with the consequent decrease in unplanned consultations, whether at primary care or at the hospital. This necessarily leads to an increase in the resolving capacity of primary care teams and an increase in the prevention of hospitalizations.

Although the role of digital technologies, as an element of support for integrated care services, is well-demonstrated, at present, we still do not have adequate digital tools that provide adequate support for collaborative work between professionals and, in turn, encourage the empowerment for self-management of patients. We understand as such, technologies: (i) compliant with the General Data Protection Regulation (GDPR), (ii) interoperable with existing health information systems, and, that (iii) facilitate the adaptive and collaborative management of chronic patients.

The present study evaluates the potential of an industry 4.0 system, Health-Circuit, based on communication technologies and intelligent collaboration, for the improvement of the management of chronic patients, with the consequent increase of the resolving capacity of the community health teams. Health-Circuit allows patients and professionals to interact, bilaterally or in groups, from various information systems and devices, regardless of their physical location. The base technology platform, Circuit, is robust (TRL 9), located in the cloud (private, mixed or public) and complies with the General Data Protection Regulation (GDPR). Circuit allows multimedia corporate communication (chat, call, video-call, file exchange, etc.) between healthcare levels, increasing coordination among professionals with the consequent improvement of health outcomes. Its potential can be increased in the future with the use of intelligent Chatbots to guide patients and professionals through complex care processes, providing decision support for personalised service selection by means of enhanced health risk assessment and patient stratification.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the SELFIE study.
* Accepting to participate in the study and sign the consent.
* In the intervention group, having a "smart phone" or "Tablet" that can support the use of the computer tool (versions of the operating systems Android or iOS compatible with the patient's application) and having an internet connection.

Exclusion Criteria:

* Physical or psychological health problems that prevent the use of the tool and that the patient does not have the help of a caregiver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Unplanned visits | 3 months
  Number of unplanned primary care and hospital visits

SECONDARY OUTCOMES:
Service utilization measures | 3 months
  number of primary care and hospital visits, number of remote resolutions and number of hospitalizations
Change in The Health Empowerment Scale | 3 months
  The instrument retained 8 items, scored on a 5 points Likert scale ranging from 5 (strongly agree) to 1 (strongly disagree). Higher scores indicate stronger level of health-related empowerment.
Change in the Fantastic Lifestyle questionnaire | 3 months
  This questionnaire contains 25 closed items that you explore nine related physical, psychological and social categories or domains to the lifestyle. It presents three response options with a numerical value of 0 to 2 for each category, and they are graded using a Likert scale, with a score of 0 to 100 points. Taking as a cut-off point the average of the qualifications proposed by the authors of the instrument five levels of qualification stratify the behavior: (<39 points = danger exists, 40 to 59 points = bad, 60 to 69 points = regular , 70 to 84 points = good, 85 to 100 points = excellent) lifestyle. The lower the score, the greater the need for change.
Equipment failures | 3 months
  Number of equipment failures according to blockage, breakage, acceleration or delay and unidentified failures
Software failures | 3 months
  Number of software failures described as slowdown in execution, information delay, command rows or information not available
Errors in execution | 3 months
  Number of errors in execution (wrong sequence action) described as omission, forward jump, backward jump, repetition, inversion or incorrect action
Number of errors due to the participant's temporary functions | 3 months
  Number of errors due to the participant's temporary functions described as forgetfulness, incorrect memory, incomplete memory, random actions, stoppage of actions, suspended task, task not completed, objective forgotten or loss of orientation
Errors due to failures in the organization | 3 months
  Number of errors due to failures in the organization described as anthropometric problems or inadequate interface
Number of participants in the study with respect to the total of potential participants | 3 months
  Number of participants in the study with respect to the total of potential participants of: i. Patients ii. Professionals
Number of entries to the application (app) per patient | 3 months
  Number of entries to the application (app) per patient
Number of contacts with clinical professionals responsible for managing the case | 3 months
  Number of contacts with clinical professionals responsible for managing the case that will be contacted through the technological tool (mHealth manager): i. Number of total contacts. ii. Number of patients who have contacted
Number of video calls | 3 months
  Number of video calls i. Number of total video calls. ii. Number of patients who have contacted via video call.
Number of patients who have accessed the conditions of use | 3 months
  Number of patients who have accessed the conditions of use
Change in Continuity of care within the healthcare system as measured by the Nijmegen Continuity of Care Questionnaire | 3 months
  It consists of four questions selected from the domain Collaboration between care of the Nijmegen Continuity of Care Questionnaire. Scored on a 5 points Likert scale ranging from 5 (strongly agree) to 1 (strongly disagree). Higher scores indicate stronger level of Collaboration between care providers from the patient's perspective.
Patient satisfaction with the mHealth tool assessed by the Net Promoter Score alongside three custom made general satisfaction. | 3 months
  The Net Promoter Score is calculated based on the answers to a single question. The result is calculated by dividing the percentage of promoters (who have a score of 9-10) minus the percentage of detractors (who have a score of 0-6). The percentage of "liabilities" (which obtained a score of 7-8) is not included in the NPS calculation. The NPS varies between -100 and +100. A positive score is considered good. The three custom made general satisfaction question is scored on a 5-point Likert scale that ranges from 0 (poor) to 10 (Good).
Professional satisfaction with the mHealth tool assessed by the Net Promoter Score alongside three custom made general satisfaction. | 3 months
  The Net Promoter Score is calculated based on the answers to a single question. The result is calculated by dividing the percentage of promoters (who have a score of 9-10) minus the percentage of detractors (who have a score of 0-6). The percentage of "liabilities" (which obtained a score of 7-8) is not included in the NPS calculation. The NPS varies between -100 and +100. A positive score is considered good. The three custom made general satisfaction question is scored on a 5-point Likert scale that ranges from 0 (poor) to 10 (Good).
Patient mHealth tool usability assessed by the System Usability Scale | 3 months
  The System Usability Scale is a 10 item questionnaire with 5 response options. Scored on a 5 points Likert scale ranging from 5 (strongly agree) to 1 (strongly disagree). Higher scores indicate stronger level of Collaboration between care providers from the patient's perspective.
Professional mHealth tool usability by the System Usability Scale | 3 months
  The System Usability Scale is a 10 item questionnaire with 5 response options. Scored on a 5 points Likert scale ranging from 5 (strongly agree) to 1 (strongly disagree). Higher scores indicate stronger level of Collaboration between care providers from the patient's perspective.
Patient mHealth experience | 3 months
  Two open questions regarding negative and positive aspects of the use of the computer tool
Professional mHealth experience | 3 months
  Two open questions regarding negative and positive aspects of the use of the computer tool
Number of clinical diagnoses in app users | 3 months
  number of high priority clinical diagnoses in app users according to CIE10 in medical history
Degree of severity of the symptom | 3 months
  Degree of severity of the symptom measured according to very mild, mild, neutral, severe or very serious
Duration of the symptom | 3 months
  Duration of the symptom expressed in hours, days or weeks
Number of professionals that the manager has contacted through the app | 3 months
  Number of professionals that the manager has contacted through the app
Number of interactions between professionals through the app | 3 months
  Number of interactions between professionals through the app
Number of solutions provided only by the manager | 3 months
  Number of solutions provided only by the manager regarding the number of total solutions
Number of solutions provided by the primary care professional | 3 months
  Number of solutions provided by the primary care professional regarding the number of total solutions
Number of solutions that has been a virtual visit | 3 months
  Number of solutions that has been a virtual visit with the primary care professional regarding the total number of solutions
Number of solutions that has been a classroom visit | 3 months
  Number of solutions that has been a classroom visit with the primary care professional regarding the total number of solutions
Number of referrals to the emergency department regarding the total number of solutions | 3 months
  Number of referrals to the emergency department regarding the total number of solutions

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Aymerich J, Hernandez C, Alonso A, Casas A, Rodriguez-Roisin R, Anto JM, Roca J. Effects of an integrated care intervention on risk factors of COPD readmission. Respir Med. 2007 Jul;101(7):1462-9. doi: 10.1016/j.rmed.2007.01.012. Epub 2007 Mar 6. PMID 17339106
- [Background] Tistad M, Lundell S, Wiklund M, Nyberg A, Holmner A, Wadell K. Usefulness and Relevance of an eHealth Tool in Supporting the Self-Management of Chronic Obstructive Pulmonary Disease: Explorative Qualitative Study of a Cocreative Process. JMIR Hum Factors. 2018 Oct 26;5(4):e10801. doi: 10.2196/10801. PMID 30368440
- [Background] Lupianez-Villanueva F, Anastasiadou D, Codagnone C, Nuno-Solinis R, Garcia-Zapirain Soto MB. Electronic Health Use in the European Union and the Effect of Multimorbidity: Cross-Sectional Survey. J Med Internet Res. 2018 May 3;20(5):e165. doi: 10.2196/jmir.7299. PMID 29724702
- [Background] Wildenbos GA, Maasri K, Jaspers M, Peute L. Older adults using a patient portal: registration and experiences, one year after implementation. Digit Health. 2018 Sep 2;4:2055207618797883. doi: 10.1177/2055207618797883. eCollection 2018 Jan-Dec. PMID 30186619
- [Background] Steele Gray C, Wodchis WP, Upshur R, Cott C, McKinstry B, Mercer S, Palen TE, Ramsay T, Thavorn K; Project Collaborators And Technology Partner, QoC Health Inc. Supporting Goal-Oriented Primary Health Care for Seniors with Complex Care Needs Using Mobile Technology: Evaluation and Implementation of the Health System Performance Research Network, Bridgepoint Electronic Patient Reported Outcome Tool. JMIR Res Protoc. 2016 Jun 24;5(2):e126. doi: 10.2196/resprot.5756. PMID 27341765
- [Background] Matui P, Wyatt JC, Pinnock H, Sheikh A, McLean S. Computer decision support systems for asthma: a systematic review. NPJ Prim Care Respir Med. 2014 May 20;24:14005. doi: 10.1038/npjpcrm.2014.5. PMID 24841952
- [Background] Leijten FRM, Struckmann V, van Ginneken E, Czypionka T, Kraus M, Reiss M, Tsiachristas A, Boland M, de Bont A, Bal R, Busse R, Rutten-van Molken M; SELFIE consortium. The SELFIE framework for integrated care for multi-morbidity: Development and description. Health Policy. 2018 Jan;122(1):12-22. doi: 10.1016/j.healthpol.2017.06.002. Epub 2017 Jun 20. PMID 28668222
- [Background] Vázquez R, Martínez M. Ministerio de Industria, Energía y Turismo Entidad Pública Empresarial Red.es Observatorio Nacional de las Telecomunicaciones y de la Sociedad de la Información [Internet]. 2016. p. 0-200. Available from: https://www.ontsi.red.es/ontsi/sites/ontsi/files/los_ciudadanos_ante_la_e-sanidad.pdf
- [Background] Reichheld FF. The one number you need to grow. Harv Bus Rev. 2003 Dec;81(12):46-54, 124. PMID 14712543
- [Result] Ramirez-Velez R, Agredo RA. [The Fantastic instrument's validity and reliability for measuring Colombian adults' life-style]. Rev Salud Publica (Bogota). 2012 Mar-Apr;14(2):226-37. doi: 10.1590/s0124-00642012000200004. Spanish. PMID 23250366
- [Result] Serrani Azcurra DJ. Elders Health Empowerment Scale: Spanish adaptation and psychometric analysis. Colomb Med (Cali). 2014 Dec 30;45(4):179-85. eCollection 2014 Oct-Dec. PMID 25767307
- [Result] Uijen AA, Schellevis FG, van den Bosch WJ, Mokkink HG, van Weel C, Schers HJ. Nijmegen Continuity Questionnaire: development and testing of a questionnaire that measures continuity of care. J Clin Epidemiol. 2011 Dec;64(12):1391-9. doi: 10.1016/j.jclinepi.2011.03.006. PMID 21689904
- [Derived] Herranz C, Martin-Moreno Banegas L, Dana Muzzio F, Siso-Almirall A, Roca J, Cano I. A Practice-Proven Adaptive Case Management Approach for Innovative Health Care Services (Health Circuit): Cluster Randomized Clinical Pilot and Descriptive Observational Study. J Med Internet Res. 2023 Jun 14;25:e47672. doi: 10.2196/47672. PMID 37314850
- See also: Digital tool — http://eu.yourcircuit.com
- See also: Measuring Usability With The System Usability Scale (SUS). Measuring Usability — http://measuringu.com/umux-lite/